CLINICAL TRIAL: NCT04862481
Title: Older Citizens During Municipality-based Rehabilitation
Brief Title: Physical Function of Older Citizens During Municipality-based Rehabilitation
Status: Completed | Type: Observational
Sponsor: University College Absalon (Other)
Collaborators: University of Southern Denmark (Other); Sundhed og Træning, Slagelse Municipality (Unknown); Danish Council for Independent Research (Other)
Responsible Party: Principal Investigator, Sanel Teljigovic, Principal Investigator, University College Absalon
Other Study IDs: SJ758; 8045-00052B (Other: Danish Council for Independent Research)
Record Dates: First submitted 2021-04-15; First posted 2021-04-28 (Actual); Last update posted 2022-03-23 (Actual); Status verified 2022-03

CONDITIONS: Aging; Rehabilitation; Frailty; Sarcopenia; Fractures, Bone; Musculoskeletal Pain; Musculoskeletal Diseases; Musculoskeletal Injury; Muscle Weakness; Weakness, Muscle
Keywords: SMFA; SF36; ICF; OLDER; REHABILITATION
MeSH Terms: conditions — Frailty; Sarcopenia; Fractures, Bone; Musculoskeletal Pain; Musculoskeletal Diseases; Muscle Weakness

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
When choosing outcomes to assess rehabilitation's effect or progress, it is essential to consider the constructs being measured and their value to the patient and the psychometric properties. Choosing an outcome that reflects all aspects of International Classification levels of Functioning, Disability and Health (ICF) is challenging, especially in heterogeneous groups. However, it is important to know the psychometric properties as this gives important knowledge on how to interpret results and, consequently, how this can inform the patient's care. The Short Musculoskeletal Function Assessment (SMFA) questionnaire can reflect differences in patients' functional status with a broad range of disorders, like for elderly citizens undergoing municipality-based rehabilitation. Nevertheless, since there is no golden standard to measure rehabilitation outcomes, construct validity needs to be established to investigate how scores of SMFA can be related to measures on all levels of ICF.

Therefore, this study has three main objectives:

1. To investigate how scores of the SMFA questionnaire are related to measures on different ICF levels
2. To describe the characteristics of older citizens starting municipality-based rehabilitation on all ICF levels
3. To investigate predictor variables of upper- and lower extremity strength

DETAILED DESCRIPTION:
The present study is a sub-study to the Randomized Controlled Trial (NCT04091308).

The present study aims to include 115 participants who will undergo measures specified in the "Outcome" section. The principal investigator of the study will conduct the testing.

ELIGIBILITY:
Inclusion Criteria:

All citizens that are referred to the health/rehabilitation center aged ≥ 65 years from Slagelse municipality will be invited to a screening interview with a physiotherapist after which the participant will be asked to join the study if not subject to one of the following exclusion criteria's:

Exclusion Criteria:

* Inability to speak or read Danish,
* Active cancer,
* Upper or lower limb amputations,
* Hypertension >180/110,
* Referred to rehabilitation primarily due to gynecological or neurological conditions (apoplexies) or surgeries where movement restrictions prohibit participating in most of the tests,
* Discouragement from a general practitioner.

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Study Population: Participants from Slagelse municipality's community-based health centre will be recruited in the period January 2021- June 2021 or until 115 men and woman have been included.
  To detect a correlation coefficient of minimum r=+/-0.3 with a significance level of 0.05 and power of 0.8 between the primary outcome SMFA and the generic health-related quality of life questionnaire SF36 a minimum of 85 participants are needed based on the Fisher's z test.
  Some studies have shown a response rate for the SMFA to be approximately 65% in cross-sectional studies, we, therefore add another 35% extra participants to the calculated sample size, resulting in a target of 115 participants to be initially included in the study.
Sampling Method: Non-Probability Sample
Enrollment: 115 (Actual)
Dates: Start 2021-01-25 (Actual); Primary Completion 2021-09-10 (Actual); Study Completion 2021-09-12 (Actual)

PRIMARY OUTCOMES:
Measure of physical functioning with Short Musculoskeletal Function Assessment (SMFA) | Baseline
  Self reported

SECONDARY OUTCOMES:
Measure in health-related quality of life with Short Form 36 (SF-36) | Baseline
  The SF-36 is a generic questionnaire that measures health-related quality of life in the past four weeks. The questionnaire consists of 36 questions which are divided into eight sub-scales and summarized in two sum scores. Higher scores indicate better health status.

OTHER OUTCOMES:
Measure of mobility with The New Mobility Score | Baseline
  The New Mobility Score assesses the patient's walking function inside, outside, and during shopping. Including whether a walking aid is used. The NMS provides a composed score of the participants' mobility. Each question is scored between 0-3 points, depending on the degree of help. The total possible score is between 0 and 9 points.
Measure of the PRISMA-7 score | Baseline
  The PRISMA-7 questionnaire is composed of seven items and is used to indicate frailty among participants - each question scores either 0 or 1 points. The total possible score is between 0 and 7 points.
Measure of the Tilburg Frailty Scale score | Baseline
  The Tilburg Frailty Scale is a questionnaire with a bio-psycho-social approach, which measures frailty. It is composed of 15 multidimensional questions, regarding the physical, psychological, and social aspects of human functioning.
  Scoring range is between 0-15 points.
Measure of pain (region of pain, intensity of pain, duration of pain), physical activity level and demographic information | Baseline
  A survey with self-formulated questions regarding name, sex, personal ID (CPR number), educational level, the region of pain the last three months (marked on a body chart), pain intensity and pain duration at the most painful body region the last three months, and physical activity level will also be collected.
Measure of weight | Baseline
  Weight will be measured in kilograms
Measure of height | Baseline
  Height will be measured in meters
Measure of blood pressure | Baseline
  Systolic and diastolic blood pressure (mmHg) will be measured using the Omron HBP 1100 blood pressure and resting heart rate monitor.
Measure of resting heart rate | Baseline
  Resting heart rate (in beats per minute) will be measured using the Omron HBP 1100 blood pressure and resting heart rate monitor.
Measure of lean body mass | Baseline
  The electrical bioimpedance device used in the present study to measure changes in body composition is the "Tanita 9MC-780U Multi Frequency Segmental Body Composition Analyzer". Lean body mass will be measured in kilograms.
Measure of fat percentage | Baseline
  The electrical bioimpedance device used in the present study to measure changes in body composition is the "Tanita 9MC-780U Multi Frequency Segmental Body Composition Analyzer". Lean body mass will be measured in kilograms.
  Fat percentage will be measured as a percentage of the total body mass.
Measure of total body water | Baseline
  The electrical bioimpedance device used in the present study to measure changes in body composition is the "Tanita 9MC-780U Multi Frequency Segmental Body Composition Analyzer". Lean body mass will be measured in kilograms.
  Total body water will be measured as percentage of the total body mass.
Measure of visceral fat | Baseline
  The electrical bioimpedance device used in the present study to measure changes in body composition is the "Tanita 9MC-780U Multi Frequency Segmental Body Composition Analyzer". Lean body mass will be measured in kilograms.
  Visceral fat will be measured on a scale ranging between 1-59. Scores above 12 indicate an unhealthy level of visceral fat.
Measure of basic metabolic rate (BMR) | Baseline
  BMR will be estimated by a bioelectrical impedance analysis device "Tanita 9MC-780U Multi Frequency Segmental Body Composition Analyze" in kilojoules.
Measure of Waist-To-Hip ratio | Baseline
  The circumference of the waist (in centimeters) will be divided with the circumference of the hip (in centimeters) to report the Waist-to-hip ratio.
Measure of maximal isometric voluntary contraction of leg extension | Baseline
  A maximal isometric voluntary contraction (in newtons) for knee extension will be performed using a strain gauge.
Measure of handgrip strength | Baseline
  The handgrip strength (in kilograms) will be measured using a hydraulic handgrip dynamometer (SAEHAN).
Measure of shoulder strength | Baseline
  The shoulder abduction strength (in kilograms) will be measured using a handheld dynamometer.
Measure of elbow strength | Baseline
  The elbow flexion and extension strength (in kilograms) will be measured using a handheld dynamometer.
Measure of leg press strength | Baseline
  Five repetitions maximum (RM) strength tests will be performed in the leg press (in kilograms) to calculate one RM.
Measure of knee extension strength | Baseline
  Five repetitions maximum (RM) strength tests will be performed in knee extension (in kilograms) to calculate one RM.
Measure of calf extension strength | Baseline
  Five repetitions maximum (RM) strength tests will be performed in the calf extension (in kilograms) to calculate one RM
Measure of gait distance with the two minutes walk test (2MWT) | Baseline
  The 2MWT will measure the distance (in meters) a person can walk in two minutes. Gaits speed will be calculated by dividing the covered distance with the time (two minutes).
Measure of heart rate before and after the two minutes walk test (2MWT) | Baseline
  Heart rate (in BPM) will be measured (using the Apple Watch serie 5) before and right after the 2MWT.
Measure of Rating Perceived Exertion using The Borg Scale before and after the two minutes walk test (2MWT) | Baseline
  The Borg Rating of Perceived Exertion 6-20 scale will be used to estimate the activity intensity before and right after the 2MWT. Higher numbers indicate higher exertion.
Measure of function using the Timed Up and Go test (TUG) | Baseline
  Time is noted (in seconds) on how long it takes to get up from a chair, walk three meters, turn around and go back to the chair and sit down again.
Measure of balance using the Tandem test | Baseline
  A measure of static balance will be performed using a Tandem test. The participants will be tested in three positions for ten seconds each (feet together, semi tandem and full tandem). Time is noted (in seconds) for how long the participant can stand in each position
Measure of balance and reaction time for upper and lower extremity | Baseline
  Measures for balance and reaction time will be collected using the "Fysiometer," and the protocols within the "Fysiometer" software will be followed.
Estimation of protein and energy intake | Baseline
  Protein and energy intake will be estimated based on 24-hour dietary recall interviews.

CONTACTS AND LOCATIONS:
Overall Officials: Sanel Teljigovic, PhD student, Principal Investigator — University College Absalon & University of Southern Denmark
Locations (1):
- Sundhed og Træning, Slagelse, Region Sjælland, Denmark

REFERENCES:
- [Derived] Teljigovic S, Dalager T, Nielsen NO, Holm L, Ejvang MB, Sjogaard G, Sogaard K, Sandal LF. Development and feasibility of a conceptual model for planning individualised physical exercise training (IPET) for older adults: a cross-sectional study. BMJ Open. 2024 Mar 5;14(3):e075726. doi: 10.1136/bmjopen-2023-075726. PMID 38448065

DOCUMENTS (1):
  • Statistical Analysis Plan (2021-12-14): https://cdn.clinicaltrials.gov/large-docs/81/NCT04862481/SAP_000.pdf